CLINICAL TRIAL: NCT00643448
Title: A Randomised, Placebo-controlled, Double-blind, Parallel-group, Multicentre, Phase IIa Study to Explore the Relationship Between QTcF Interval at First Dose (Loading Dose) and at Steady State After Treatment With AZD1305 Extended-release Tablets or Placebo When Given to Patients With Documented AF
Brief Title: Explorative Study of AZD1305 in Atrial Fibrillation Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3190C00019; 2007-007058-79
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2011-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD1305 loading dose 250 mg + 125 mg (Experimental): Tablets
  Interventions: Drug: AZD1305
- AZD1305 loading dose 500 mg + placebo (Experimental): Tablets
  Interventions: Drug: AZD1305
- Placebo corresponding to AZD1305 loading dose (Placebo Comparator): Tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1305 — AZD1305 loading dose 250 mg + 125 mg evening dose on Study Day 1, maintenance dose 125 mg twice daily from Study Day 2
  Arms: AZD1305 loading dose 250 mg + 125 mg
Drug: AZD1305 — AZD1305 loading dose 500 mg + placebo evening dose on Study Day 1, maintenance dose 125 mg twice daily from Study Day 2
  Arms: AZD1305 loading dose 500 mg + placebo
Drug: Placebo — Placebo corresponding to AZD1305 loading dose + evening dose on Study Day 1, maintenance dose twice daily from Study Day 2
  Arms: Placebo corresponding to AZD1305 loading dose

SUMMARY:
Explorative study in Atrial Fibrillation patients to assess Safety and Pharmacokinetics at initiation of treatment and at steady state

ELIGIBILITY:
Inclusion Criteria:

* Documented Atrial Fibrillation but in stable SR for at least 2 h and a maximum of 28 days.
* Sinus rhythm at randomisation

Exclusion Criteria:

* Haemodynamically unstable condition as judged by the Investigator, systolic BP <100 mmHg or >180 mmHg, or diastolic BP >105 mmHg at randomisation
* Personal or family history of Torsades de Pointes (TdP), any other polymorphic ventricular tachycardia (PVT), sustained ventricular tachycardia, long QT syndrome and/or Brugada syndrome
* Sinus bradycardia (<50 beats per minute (bpm)) at randomisation
* QTc (Fridericia, QTcF ) >450 ms measured in sinus rhythm at randomisation,
* Serum potassium below 3.8 or above 5.0 mmol/L or plasma potassium below 3.6 or above 5.0 mmol/L
* QRS duration >120 ms at randomisation
* Use of any antiarrhythmic drug class I and/or III, digitalis glycoside, QT prolonging drug and/or drug that inhibits CYP3A4, as well as St John's Worth

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egstrup, Principal Investigator — Svendborg Sygehus, Forsknings-og udviklingsafd.
Locations (18):
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Hvidovre
  - Research Site, Silkeborg
  - Research Site, Svendborg
- Norway (3):
  - Research Site, Oslo
  - Research Site, Rud
  - Research Site, Tynset
- Poland (2):
  - Research Site, Bytom
  - Research Site, Warsaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Slovakia (4):
  - Research Site, Košice
  - Research Site, Nitra
  - Research Site, Nové Zámky
  - Research Site, Rimavská Sobota
- Research Site, Gothenburg, Sweden

REFERENCES:
- [Derived] Egstrup K, Bergfeldt L, Duris T, Gullestad L, Kochmanski M, Kusnierz B, Nielsen T, Sawicki S, Aunes-Jansson M, Edvardsson N, Frison L, Johansson S, Berggren A. QT response after a test dose and during maintenance therapy with AZD1305 in patients with atrial fibrillation: a double-blind, randomized, placebo-controlled trial. Am J Cardiovasc Drugs. 2011 Jun 1;11(3):199-208. doi: 10.2165/11591750-000000000-00000. PMID 21619383

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients will attend a pre-entry Visit 3-28 days before the planned randomisation. At this Visit, the Investigator ensures that a signed Informed Consent Form has been obtained before any study specific procedures are conducted. Patients who have given their consent to participate in the study will then undergo a full clinical assessment
Groups:
- AZD1305 Group A: AZD1305 group A loading dose 250 mg + 125 mg evening dose on Study Day 1, maintenance dose 125 mg twice daily from Study Day 2
- AZD1305 Group B: AZD1305 loading dose 500 mg + placebo evening dose on Study Day 1, maintenance dose 125 mg twice daily from Study Day 2
Period: Overall Study
Arm/Group | AZD1305 Group A | AZD1305 Group B | Placebo
Started | 21 | 22 | 22
Completed | 17 | 17 | 16
Not Completed | 4 | 5 | 6
Not completed — Lack of Efficacy | 2 | 0 | 4
Not completed — Adverse Event | 2 | 2 | 2
Not completed — QTcF>550 ms | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1305 Group A | AZD1305 Group B | Placebo | Total
Number analyzed (Participants) | 21 | 22 | 22 | 65
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age (years) | 65 (10) | 64 (10) | 64 (9) | 64.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 8 | 26
  Male | 13 | 12 | 14 | 39

OUTCOME MEASURES:

1. Primary Outcome: Maximum QTcF
Description: Maximum of all QTcF values obtained for any given patient from randomisation until the intended end of the study drug period, day 10.
Time Frame: During treatment days 2-10
Measure: Mean (Full Range); unit: ms
Groups:
- AZD1305 Group A and AZD1305 Group B: AZD1305 group A loading dose 250 mg + 125 mg evening dose on Study Day 1, maintenance dose 125 mg twice daily from Study Day 2 AZD1305 Group B loading dose 500 mg + placebo evening dose on Study Day 1, maintenance dose 125 mg twice daily from Study Day 2
Arm/Group | AZD1305 Group A and AZD1305 Group B | Placebo
Number analyzed (Participants) | 21 | 22
ms | 461 (417) [417 to 536] | 427 (383) [383 to 465]

2. Secondary Outcome: Adverse Events (AE)
Description: Number of patients who had at least one AE according to the definition in the study protocol
Time Frame: During treatment days 2-10
Measure: Number; unit: Participants
Arm/Group | AZD1305 Group A and AZD1305 Group B | Placebo
Number analyzed (Participants) | 43 | 21
Participants | 22 | 13

3. Secondary Outcome: Estimated Cmax (Maximum Plasma Concentration) (PK Modeling) at Steady-state
Description: Population PK model parameter estimates derived from plasma concentrations of AZD1305
Time Frame: During treatment days 1-10
Measure: Mean (Full Range); unit: μmol/L
Arm/Group | AZD1305 Group A | AZD1305 Group B | Placebo
Number analyzed (Participants) | 17 | 17 | 0
μmol/L | 0.41 (0.17) [0.17 to 0.83] | 0.45 (0.24) [0.24 to 0.84] |

4. Secondary Outcome: Compliance With Trans Telephonic Monitoring (TTM)
Description: Percentage of twice daily TTM recordings (individual compliance) transmitted and available for analysis
Time Frame: During treatment days 1-10
Measure: Mean (Full Range); unit: Percentage of recordings analysed
Arm/Group | AZD1305 Group A | AZD1305 Group B | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Percentage of recordings analysed | 97.4 (80) [80 to 100] | 96.4 (68.2) [68.2 to 100] | 98.3 (72.7) [72.7 to 100]

ADVERSE EVENTS:
Arm/Group | AZD1305 Group A | AZD1305 Group B | Placebo
Serious Adverse Events (participants affected / at risk) | 0 | 3 | 0
Other Adverse Events (participants affected / at risk) | 10 | 12 | 9
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | AZD1305 Group A | AZD1305 Group B | Placebo
Ventricular Bigeminy (Cardiac disorders) | 0/21 | 1/22 | 0/22
Polymorphic Ventricular Tachycardia (Cardiac disorders) | 0/21 | 1/22 | 0/22
Neutropenia (Blood and lymphatic system disorders) | 0/21 | 1/22 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | AZD1305 Group A | AZD1305 Group B | Placebo
Atrial Fibrillation (Cardiac disorders) | 1/21 | 0/22 | 2/22
Bradycardia (Cardiac disorders) | 1/21 | 2/22 | 1/22
Palpitation (Cardiac disorders) | 2/21 | 1/22 | 3/22
Nausea (General disorders) | 2/21 | 1/22 | 2/22
Application Site Reaction (General disorders) | 2/21 | 3/22 | 0/22
Oedema Peripheral (General disorders) | 2/21 | 0/22 | 0/22
Qt Interval Prolonged (General disorders) | 0/21 | 3/22 | 0/22
Dizziness (Nervous system disorders) | 2/21 | 4/22 | 0/22
Headache (Nervous system disorders) | 4/21 | 4/22 | 2/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less